CLINICAL TRIAL: NCT02373189
Title: Bright Light Treatment At Home To Manage Chronic Pain In U.S. Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13082603; R34AT008347 (NIH)
Record Dates: First submitted 2015-02-16; First posted 2015-02-26 (Estimated); Results first posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bright light (Experimental): Participants received morning bright light.
  Interventions: Device: Bright light

INTERVENTIONS:
Device: Bright light — The purpose of this R34 Pilot and Feasibility study is to develop a morning bright light treatment to help manage chronic pain and improve PTSD symptoms, mood, and sleep in US veterans. Veterans will have 7 baseline days at home, followed by a baseline pain sensitivity assessment and baseline home circadian phase assessment (dim light melatonin onset). Following an instructional home visit, patients will then self-administer morning bright light treatment for 6 days, followed by reassessments of pain sensitivity and home circadian phase. This will be repeated after a further 7 days of morning bright light treatment. The Patient Reported Outcomes Measurement Information System (PROMIS) will also be administered at every lab visit. Additionally, pain and mood (electronic diaries) and sleep (wrist actigraphy) will be assessed daily throughout baseline and treatment. Pain, mood and sleep will also be self-reported daily during a 1 month follow up after cessation of light treatment.

SUMMARY:
Nearly 50% of U.S. veterans report they experience pain on a regular basis. This chronic pain often co-occurs with other disorders including post-traumatic stress disorder (PTSD), depression, anxiety and insomnia. A common approach to treating chronic pain is opioid analgesics, which are not always effective, and increasingly associated with abuse and misuse. Thus, there is an urgent need to develop readily available, safe, and practical complementary nonpharmacological approaches to manage chronic pain in U.S. veterans. Chronic pain is a multidimensional phenomenon, inter-related with many factors, including negative mood and poor sleep. The central circadian clock, in the suprachiasmatic nucleus in the hypothalamus, is well recognized to regulate both mood and sleep, and even small delays (shifts later) in circadian/sleep timing are associated with depression and disrupted sleep. These results suggests that later circadian/sleep timing may be a modifiable risk factor for pain. Thus, a self-administered morning bright light treatment at home may be a potentially efficacious adjunctive strategy for managing chronic pain. This R34 grant will develop a morning bright light treatment to help manage chronic pain and improve PTSD symptoms, depression, anxiety and sleep in U.S. veterans. Patients will have 7 baseline days at home, followed by a baseline pain sensitivity assessment and home circadian phase assessment (dim light melatonin onset). Following an instructional home visit, patients will then self-administer morning bright light treatment for 6 days, followed by reassessments of pain sensitivity and circadian phase. Assessments will be repeated after another 7 days of morning bright light treatment. Pain, mood and sleep (wrist actigraphy) will be assessed daily throughout baseline and treatment. Pain, mood and sleep will also be rated by veterans daily during a 1 month follow up after cessation of light treatment. This study will determine the feasibility, acceptability and efficacy of bright light treatment in a sample of U.S. veterans experiencing chronic low back pain.

DETAILED DESCRIPTION:
Almost 50% of U.S. veterans report they experience pain on a regular basis. This chronic pain often co-occurs with other disorders including post-traumatic stress disorder (PTSD), depression, anxiety and insomnia. A common approach to treating chronic pain is opioid analgesics, which are not always effective, and increasingly associated with abuse and misuse. Thus, there is an urgent need to develop readily available, safe, and practical complementary nonpharmacological approaches to manage chronic pain in U.S. veterans. Chronic pain is a multidimensional phenomenon, inter-related with many factors, including negative mood and poor sleep. The central circadian clock, in the suprachiasmatic nucleus in the hypothalamus, is well recognized to regulate both mood and sleep, and even small delays (shifts later) in circadian/sleep timing are associated with depression and disrupted sleep. These results suggests that later circadian/sleep timing may be a modifiable risk factor for pain. Thus, a self-administered morning bright light treatment at home may be a potentially efficacious adjunctive strategy for managing chronic pain. This R34 grant will develop a morning bright light treatment to help manage chronic pain and improve PTSD symptoms, depression, anxiety and sleep in U.S. veterans. Patients will have 7 baseline days at home, followed by a baseline pain sensitivity assessment and home circadian phase assessment (dim light melatonin onset). Following an instructional home visit, patients will then self-administer morning bright light treatment for 6 days, followed by reassessments of pain sensitivity and circadian phase. Assessments will be repeated after another 7 days of morning bright light treatment. Pain, mood and sleep (wrist actigraphy) will be assessed daily throughout baseline and treatment. Pain, mood and sleep will also be rated by veterans daily during a 1 month follow up after cessation of light treatment. This study will determine the feasibility, acceptability and efficacy of bright light treatment in a sample of U.S. veterans experiencing chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. U.S. veteran
2. musculoskeletal pain of the lower back and/or leg pain stemming from degenerative disk disease, spinal stenosis, or disk herniation (radiculopathy subcategory), or muscular or ligamentous strain (chronic myofascial pain subcategory) verified with written confirmation from physician/medical record
3. age between 18 and 70 years
4. live within 1.5 hours drive of Rush University Medical Center

Exclusion Criteria:

1. inability to understand English well enough to complete questionnaires or to participate;
2. unable to travel to the lab

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen J Burgess, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Trial of Bright Light Treatment for Chronic Pain: Bright light: The purpose of this R34 Pilot and Feasibility study is to develop a morning bright light treatment to help manage chronic pain and improve PTSD symptoms, mood, and sleep in US veterans. Veterans will have 7 baseline days at home, followed by a baseline pain sensitivity assessment and baseline home circadian phase assessment (dim light melatonin onset). Following an instructional home visit, patients will then self-administer morning bright light treatment for 6 days, followed by reassessments of pain sensitivity and home circadian phase. This will be repeated after a further 7 days of morning bright light treatment. The Patient Reported Outcomes Measurement Information System (PROMIS) will also be administered at every lab visit. Additionally, pain and mood (electronic diaries) and sleep (wrist actigraphy) will be assessed daily throughout baseline and treatment. Pain, mood and sleep will also be self-reported daily during a 1 month follow up after cessation of light treatment.
Period: Overall Study
Arm/Group | Open Trial of Bright Light Treatment for Chronic Pain
Started | 37
Completed | 25
Not Completed | 12

BASELINE CHARACTERISTICS:
Population: US military veterans with chronic low back pain
Arm/Group | Open Trial of Bright Light Treatment for Chronic Pain
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] — Demographic information on average age of participants. Lowest age available for each participant 18 and highest age 65. We describe the mean age of our participants. There is no subscale data or better or worse for this description.
  years | 48.4 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Information gathered on two different sexes of our participants. Male and Female descriptors used with totals listed for percentages of each category. This is not a scale measurement just direct information on participants. No better or worse outcomes for this and no subscale.
  Participants
    Female: Female | 10
    Female: Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants] — Breakout of different race descriptors for participants. There is no subscale and no better or worse metrics used. Use of commonly used race descriptors for participants used.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 22
    White | 13
    More than one race | 2
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Measurement to determine different locations of participants per country location. There is no subscale and no better or worse scale.
  participants
    United States | 37
pain intensity [Mean (Standard Deviation); unit: units on a scale] — PROMIS Pain Intensity Scale. The first two items in the Pain Intensity item bank assess pain intensity utilizing a 7-day recall period (items include the phrase "the past 7 days") while the last item asks patient to rate their pain intensity "right now." The Pain Intensity instrument is available for adults (ages 18+). A Numerical Rating Scale, patients are asked to circle the number between 0 and 100 that fits best to their pain intensity. "0" represents 'no pain at all' whereas "100" represents 'the worst pain ever possible'. Likert scale used 0-100 with median at 50.
  units on a scale | 47.02 (6)

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Outcomes Measurement Information System Pain Intensity
Description: How intense is the pain? 0-100 Likert Scale. 0 = no pain; 100 = worst pain
Time Frame: 1 day
Population: US military veterans
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Trial of Bright Light Treatment for Chronic Pain
Number analyzed (Participants) | 25
units on a scale | 48.84 (6.30)
Statistical Analysis 1: Comparison: Open Trial of Bright Light Treatment for Chronic Pain; Test type: Superiority; p = 0.05, paired t-test — The P-value indicated above is calculated; means at pre and post treatment were compared within subject

2. Secondary Outcome: Pain Tolerance
Description: Laboratory testing. Subject placed hand in ice water until discomfort became intolerable. Elapsed time between immersion and removal of hand in seconds was defined as "tolerance."
Time Frame: 0 - 5 minutes
Population: US military veterans
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Open Trial of Bright Light Treatment for Chronic Pain
Number analyzed (Participants) | 25
seconds | 187.88 (160.13)
Statistical Analysis 1: Comparison: Open Trial of Bright Light Treatment for Chronic Pain; Test type: Superiority; p = 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 day
Description: Procedures were deemed low risk.
Arm/Group | Open Trial of Bright Light Treatment for Chronic Pain
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT02373189/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT02373189/SAP_001.pdf
  • Informed Consent Form (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT02373189/ICF_002.pdf